CLINICAL TRIAL: NCT04688151
Title: Phase Ib, Multi-center Study of Combining Rituximab, Acalabrutinib, and Durvalumab (RAD) in Primary Central Nervous System Lymphoma.
Brief Title: Rituximab, Acalabrutinib, and Durvalumab (RAD) in Primary CNS Lymphoma.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); National Cheng-Kung University Hospital (Other); China Medical University Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2420
Record Dates: First submitted 2020-12-08; First posted 2020-12-29 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-04

CONDITIONS: Primary Central Nervous System Lymphoma (PCNSL)
MeSH Terms: interventions — Rituximab; acalabrutinib; durvalumab

STUDY DESIGN:
Intervention Model Description: Dose level 1,Dose level 2,3+3 design in the dose escalation.
Masking Description: This study will use the 3+3 design in the dose escalation phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose level 1,Dose level 2 (Experimental): Dose level 1 Rituximab 375mg/m2 infusion once every 4 weeks for 8 cycles Acalabrutinib 100mg PO once every day Durvalumab 1500mg infusion once every 4 weeks Dose level 2 Rituximab 375mg/m2 infusion once every 4 weeks for 8 cycles Acalabrutinib 100mg PO twice every day Durvalumab 1500mg infusion once every 4 weeks
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Dose level 1:Rituximab 375mg/m2 infusion once every 4 weeks for 8 cycles Acalabrutinib 100mg PO once every day Durvalumab 1500mg infusion once every 4 weeks Dose level 2:Rituximab 375mg/m2 infusion once every 4 weeks for 8 cycles Acalabrutinib 100mg PO twice every day Durvalumab 1500mg infusion once every 4 weeks Expansion:Determined by the result of the dose escalation phase
  Other Names: Acalabrutinib; Durvalumab

SUMMARY:
To evaluate the safety and tolerability and determine the recommended phase 2/phase 3 dose of RAD regimen in PCNSL

DETAILED DESCRIPTION:
Target subject population Male and female patients with PCNSL who have failed to achieve a response or who have relapsed after prior therapy (R/R) or who are treatment naïve but are not candidates of standard high-dose methotrexate-based induction chemotherapy. Patients are not to have been previously treated with immune checkpoint inhibitors or Bruton tyrosine kinase (BTK) inhibitors; prior treatment with rituximab is allowed.

Duration of treatment Rituximab will be administered for up to 8 cycles or until intolerance or excessive toxicities relevant to the trial therapy, or withdrawal of consents; acalabrutinib and durvalumab will be continued until disease progression, intolerance, or excessive toxicities relevant to the trial therapy, or withdrawal of consents.

Investigational product, dosage, and mode of administration Dose level 1 Rituximab 375mg/m2 infusion once every 4 weeks for 8 cycles Acalabrutinib 100mg PO once every day Durvalumab 1500mg infusion once every 4 weeks Dose level 2 Rituximab 375mg/m2 infusion once every 4 weeks for 8 cycles Acalabrutinib 100mg PO twice every day Durvalumab 1500mg infusion once every 4 weeks Expansion Determined by the result of the dose escalation phase Statistical methods

This study will use the 3+3 design in the dose escalation phase. Analyses will be primarily descriptive in nature; no formal statistical hypothesis testing will be performed. The populations used for analysis will include the following:

Safety analysis set: patients who receive at least 1 dose of anyone of the study drugs will be used for safety analyses.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, 20 years of age or older.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 3.
* Histologically or cytologically proven diagnosis of primary CNS lymphomas of large B-cell type in one of the following clinical status:
* Fail to achieve optimal response (CR or PR) after at least one prior therapy with all the toxicities recovered to grade 1 or less from the prior therapy.
* Has confirmed disease relapse or disease progression after at least one prior therapy with all the toxicities recovery to grade 1 or less from the prior therapy.
* Intolerable to the prior therapy because of toxicities with all the toxicities recovery to grade 1 or less from the prior therapy.
* Treatment naïve but unable or not willing to receive high-dose methotrexate-based induction chemotherapy.
* Have at least one measurable brain parenchymal lesion that can be measured by brain MR or CT images.
* Have adequate organ functions as defined by the following criteria:
* Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≦3 x upper limit of normal (ULN).
* Total serum bilirubin ≦2 x ULN (except for Gilbert's syndrome)
* Absolute neutrophil count (ANC) ≧1,000/mL; Platelets ≧50,000/mL; Hemoglobin≧8.0 g/dL.
* Serum creatinine ≦2.0 x ULN.
* Prothrombin time/International normalized ratio (PT/INR) ≦2.0 x ULN and partial thromboplastin time (PTT) ≦2.0 x ULN.
* Any major surgery must have been completed at least 4 weeks prior to study entry. Any prior therapies, including chemotherapy, rituximab, or high dose or high potency corticosteroids intended to treat lymphoma (dose higher than 100 mg hydrocortisone per day or equivalent potency), must have been completed at least 2 weeks prior to the study entry. However, low-dose, low-potency steroids (ie, up to 100 mg hydrocortisone per day or equivalent potency) may be used prior to the initiation of the trial therapy for the relief of lymphoma-related symptoms. Non-regular steroid administration for premedication purpose are allowed (refer to section 7.7). Any prior radiation performed with curative (i.e., not only palliative) intent or minor surgeries/procedures must have been completed at least 2 weeks prior to the initiation of study medication. Palliative radiation (≤10 fractions) must have been completed 48 hours prior the start of the trial therapy commencing. Any acute toxicity must have been recovered to grade 1 (except alopecia).
* Life expectancy ≥12 weeks in the opinion of the investigator.
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrolment.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, tissue, CSF, and blood sample collections for explorative objectives and other study procedures.
* Male and female patients of childbearing potential must agree to use a highly effective method of contraception throughout the study and for 12 months after the last dose of RAD or at least 2 days after the last dose of aclabrutinib monotherapy, if the patient receives acalabrutinib monotherapy for greater than 12 months after the last dose of RAD administration. A patient is of childbearing potential if he/she is biologically capable of having children and is sexually active

Exclusion Criteria:

* Diagnosis with secondary CNS lymphoma, i.e. systemic lymphoma with CNS involvement or relapse, or diagnosis with PCNSL but with other non-CNS, systemic involvement.
* Active or uncontrolled autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:
* Patients with vitiligo or alopecia.
* Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement.
* Patients with any chronic skin condition that does not require systemic therapy.
* Patients with other autoimmune or inflammatory disorders that are not active in the last 2 years may be included.
* Patients with celiac disease controlled by diet alone.
* History of another primary malignancy except for:
* Malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of the trial therapy and of low potential risk for recurrence.
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
* Adequately treated carcinoma in situ without evidence of disease.
* Has positive HBV surface antigen (HBsAg) result. Patients who are negative for HBsAg but are positive for anti-HBc antibody are allowed to be enrolled if their HBV-DNA test are negative.
* Has positive HCV-RNA result.
* Has positive anti-human immunodeficiency virus (HIV)-1/2 antibody test results.
* Prior history of anaphylaxis or severe allergic reactions to anyone of the study drugs or the excipients.
* Prior exposures to checkpoint inhibitors or BTK inhibitors.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of the trial therapy. Note: Patients, if enrolled, should not receive live vaccine while receiving the trial therapy and up to 30 days after the last dose of the trial therapy.
* Has active infection, as ascertained by the investigator, which might result in extra-risk of toxicities with the administration of the trial therapy.
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study. Participation in another clinical study with the last investigational therapy administration must be finished at least 4 weeks ago before initiating the current RAD trial therapy.
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
* Previous allogeneic hematopoietic stem cell transplant.
* Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site).
* Known history of drug or alcohol abuse within 2 years of screening.
* Any concomitant medications that are known to be associated with Torsades de Pointes or requires treatments with strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers.
* For women only - currently pregnant (confirmed with positive pregnancy test) or breastfeeding.
* Has history of arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which is symptomatic or requires treatment (CTCAE Grade 3 to 4), symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Subjects with atrial fibrillation controlled by medication are permitted.
* Has current active bleeding disorders or has history of bleeding diathesis.
* Requires warfarin or Vit. K antagonist administration.
* Has history of myocardial infarction.
* Has recent history of vascular stroke or CNS haemorrhagic stroke within 6 months.
* Has confirmed or suspected progressive multifocal leukoencephalopathy
* Has difficulty in swallowing oral medications or has significant gastrointestinal diseases that would limit the absorption of oral medications.
* Has clinically significant cardiac diseases as defined by New York Association Classification class 3 or 4.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
MTD of acalabrutinib | From date of registration until the date of definition of MTD of first documented progression or date of death from any cause, whichever came first, assessed up to 28 weeks.
  Dose-limiting toxicity (DLT) patients will be enrolled in cohort of 2 to receive escalating dose of acalabrutinib at two dose levels (level I 100mg PO once , level II 100mg PO twice every day) or more of defined events

SECONDARY OUTCOMES:
Tumor response | From date of registration until the date of definition of MTD of first documented progression or date of death from any cause, whichever came first, assessed up to 28 weeks.
  Efficacy evaluation: objective tumor response according to International PCNSL Collaborative Group Guidelinefor Response Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Shang-Ju Wu, M.D, Principal Investigator — National Taiwan University Hospital, Taipei, Taiwan; Su-Peng Yeh, M.D, Principal Investigator — China Medical University Hospital; Kwang-Yu Chang, M.D, Principal Investigator — National Cheng Kung University Hospital,Taiwan; Ming Chung Wang, M.D, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Shang-Ju Wu, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No